CLINICAL TRIAL: NCT06587542
Title: Comparison of the Response and Pathomechanism of Purified Tuberculin Unit Protein Injection Therapy for Anogenital Warts with and Without HIV Infection
Brief Title: Effectivity of Protein Purified Derivative Treatment for Anogenital Warts in HIV Patient
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DV-202407.01
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Anogenital Warts; HIV Infection; Tuberculin Purified Protein Derivative
Keywords: anogenital warts; HIV infection; tuberculin purified protein derivative
MeSH Terms: conditions — Condylomata Acuminata; HIV Infections

STUDY DESIGN:
Intervention Model Description: Patients having anogenital warts will be divided into 2 groups, i.e. HIV and non-HIV groups. Both groups will receive a single injection of tuberculin PPD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIV-positive patients with anogenital warts (Experimental): Injection of protein purified derivative
  Interventions: Other: Injection of protein purified derivative
- HIV-negative patients with anogenital warts (Experimental)
  Interventions: Other: Injection of protein purified derivative

INTERVENTIONS:
Other: Injection of protein purified derivative — Injection of purified protein derivative for anogenital warts in HIV and non HIV patient, on the largest lesion

SUMMARY:
Warts are a common viral infection of the skin and are prevalent throughout the world, with an overall prevalence in the United States estimated at 2-20%. The incidence of anogenital warts occurs more frequently in HIV-infected patients, with a seven-fold increase in risk compared to patients without HIV infection. Available treatments for anogenital warts can only reduce, but cannot eradicate, HPV infection. There are many therapeutic options for treating anogenital warts, but none can prevent recurrence. Immunotherapy has become one of the best therapeutic options for warts caused by HPV infection because it increases the immune response to HPV infection, resulting in remission, both in lesions that receive direct and indirect intralesional therapy. Immunotherapy, acts as a basic principle to enhance cell-mediated immunity for wart clearance. Apart from low recurrence, regression in immunotherapy for warts due to HPV infection generally occurs without cicatrices, so it is a consideration in choosing therapy, including anogenital warts. Various types of immunotherapy have been used, one of which is purified protein derivative, which can be used as an alternative therapy option for anogenital warts. In a previous case report, even though an HIV patient had an abnormal immune system, tuberculin protein purified derivative therapy, immunotherapy provided a significant clinical response in the form of a reduction in lesion size, compared to patients who were not given therapy. Research regarding the comparison of the response to tuberculin protein purified derivative therapy in anogenital warts patients with and without HIV infection has never been reported. Therefore, researchers are interested in examining the comparison of the response to tuberculin purified protein derivative therapy in anogenital warts patients between those with and without HIV infection and knowing the comparison of local and systemic cytokine changes when administering anogenital wart therapy with tuberculin protein purified derivative between those with and without HIV infection.

DETAILED DESCRIPTION:
Research Design Research on the response to administration of intralesional PPD-2TU therapy in warts to changes in levels of various cytokines locally and systemically.

Data, Data Collection Techniques and Data Sources The data used is primary data. Primary data is the result of examination anogenital warts patients who were then given PP2-TU therapy at varying doses, blood serum and histopathological preparations are taken before injection and 3 weeks after the injection.

Sample Taking/Selection The research sample was anogenital warts patients who were treated at the Infection Polyclinic Sexually Transmitted Hospital Dr. Hasan Sadikin Bandung, using consecutive sampling for each group, 15 anogenital warts patients with and 15 patient without HIV infection were given purified protein derivative injection.

Data Validity and Reliability The validity of laboratory examination data can be guaranteed due to inspection. Laboratory work is carried out in the clinical pathology and anatomical pathology laboratories of the Hospital Dr Hasan Sadikin who has international standards.

Independent variable: Patients with anogenital warts Dependent variables: Clinical response, levels of IFN-α, IFN-γ, and IL-2 in the blood and tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Anogenital warts whose diagnosis is made based on anamnesis and physical examination, before receiving intralesional purified protein derivative injection therapy.
2. All stored biological materials that have been previously taken through tissue from anogenital warts patients whose diagnosis was confirmed based on history and physical examination, 3 weeks after receiving the first intralesional purified protein derivative injection therapy.

Exclusion Criteria:

* 1. With a history of allergies to purified protein derivative, generalized dermatitis, asthma and skin allergies 2. Currently taking immunosuppressant or immunomodulatory drugs based on the history and clinical examination.

  3. Have an immunodeficiency disease based on anamnesis and clinical examination, except for HIV based on anamnesis, clinical examination and serological examination (anti-HIV).

  4. Have a history of suffering from malignancy based on history and clinical examination.

  5. Infected with tuberculosis based on history, clinical examination and chest radiography.

  6. Infected with other STIs based on history, clinical examination, and serological examination (venereal disease research laboratory (VDRL), Treponema pallidum hemagglutination assay (TPHA), and Hepatitis B surface antigen (HBsAg)).

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
clinical improvement | 3 weeks after treatment
  defined as the reduced in number which describe in number and size which describe in cm cubic of volume which obtained by measuring the length times width times height of the anogenital warts lesion

SECONDARY OUTCOMES:
cytokine change in blood and tissue | 3 weeks after treatment
  the cytokine change will be measure using ELISA for detection int the blood specimen, while cytokine change in the tissue sample will be measure with mRNA expression using PCR

IPD SHARING:
Plan to Share IPD: No
Its need the Indonesian goverment clearance for do so

REFERENCES:
- [Background] Achdiat PA, Widjaja S, Suwarsa O, Dwiyana RF, Hindritiani R, Sutedja E, Gunawan H, Usman HA, Rianty F, Maharani RH. Effectiveness and safety of tuberculin purified protein derivative for the treatment of anogenital warts in patients with human immunodeficiency virus. Dermatol Reports. 2024 Jan 30;16(3):9754. doi: 10.4081/dr.2024.9754. eCollection 2024 Sep 2. PMID 39635572